CLINICAL TRIAL: NCT04390802
Title: A Pilot Study of 5-Aminolevulinic Acid (5-ALA) to Enhance Visualization of Pituitary Adenomas
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: NX Development Corp (Industry)
Responsible Party: Principal Investigator, Pamela Stuart Jones, Assistant Professor of Neurosurgery, Massachusetts General Hospital
Other Study IDs: 2019P003509
Record Dates: First submitted 2020-04-28; First posted 2020-05-18 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: 5-aminolevulinic acid — Study participants who are deemed surgical candidates for management of their pituitary lesion will drink 20mg/kg 5-ALA 2-4 hours preoperatively. They will then be taken to the operation room and undergo general anesthesia. Intraoperative blood draw may occur from lines places for anesthesia purposes at any time during the operation. In alignment with the neurosurgeon's practice and discretion, the sella will be accessed and opened. During the surgical exploration of the sella, the surgeon will attempt to identify the pituitary mass. The location of the tumor will be assessed using the blue-light filtered microscope or endoscope. These steps will be documented photographically during the operation. A biopsy of the fluorescent region will be taken to confirm pituitary adenoma histopathology. The tumor will then be maximally resected. The tumor sample will be used for further clinical testing as part of the patient's routine care.

SUMMARY:
5-Aminolevulinic Acid (5-ALA) was approved by the FDA as an intraoperative optical imaging agent in patients with suspected high-grade gliomas (HGGs) in 2017. The investigators plan to administer 5-ALA to patients with pituitary tumors to demonstrate whether it can be used as an intraoperative optical imaging agent for this pathology. Overall, this pilot study will afford the overall opportunity to improve surgical management and advancement of the science of neurological and neuroendocrine disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-functioning pituitary adenomas who require surgical intervention, as deemed appropriate by a neurosurgeon, either due to size criteria, observed growth in lesion on MRI, and/or for alleviation of the symptoms of mass effect.
* Patients with functional pituitary adenomas, including prolactinomas, growth-hormone secreting adenomas, and ACTH-secreting adenomas, where surgery is recommended for biochemical control. Patients with symptoms of Cushing's Disease and centralization of ACTH on IPSS without imaging-confirmed lesions will be included in the study.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to aminolevulinic acid (ALA). Patients should refrain from use of other potential phototoxic substances (e.g. tetracyclines, sulfonamides, fluoroquinolones, hypericin extracts) for 72 hours.
* Personal or family history of porphyria.
* Uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 5-ALA breastfeeding should be discontinued if the mother is treated with 5-aminolevulinic acid.
* Women who are pregnant or become pregnant will be excluded from the trial as it is unknown if aminolevulinic acid (ALA) is teratogenic or has abortifacient effects.
* Prior history of GI perforation, diverticulitis, and/or peptic ulcer disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will study patients with pituitary macroadenomas who require surgical intervention, as deemed appropriate by a neurosurgeon, either due to size criteria, observed growth in lesion on MRI, and/or for alleviation of the symptoms of mass effect. The investigators will also study patients with functional pituitary adenomas, including prolactinomas, growth-hormone secreting adenomas, and ACTH-secreting adenomas, where surgery is recommended for biochemical control.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with intraoperative observed fluorescence of pituitary tumor | through study completion, an average of 3 months
  Under blue light exposure of tumor, the investigators will document whether red fluorescence is seen (+ fluorescence) or not seen (- fluorescence). These will be categorized as a binary finding. If fluorescence is seen, the surgeon will biopsy this area to confirm that fluorescent tissue is consistent with pituitary adenoma by histopathology.

SECONDARY OUTCOMES:
Differences in presence of fluorescence based on hormone receptor staining of the pituitary adenoma | through study completion, an average of 3 months
  If possible, the investigators will report differences in presence and degree of fluorescence between different types of pituitary adenomas based on their hormone receptor staining status by immunohistochemistry.